CLINICAL TRIAL: NCT06323408
Title: Prospective Collection of Clinical and Imaging Data, Radiotherapy Planning and Biomaterials for Integrated Analysis of Therapy Response and Resistance and Detection of Molecular Targets in Adolescents and Young Adults With CNS Tumors
Brief Title: Integrated Analysis of Therapy Response and Resistence in Embryonal Tumors and Gliomas
Acronym: BZKF-AYA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Peter Hau, Prof., University Hospital Regensburg
Other Study IDs: BZKF-AYA_1.0
Record Dates: First submitted 2024-03-01; First posted 2024-03-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Glioma, Malignant; Embryonal Tumor; Medulloblastoma; Ependymoma
MeSH Terms: conditions — Glioma; Neoplasms, Germ Cell and Embryonal; Medulloblastoma; Ependymoma | interventions — Histocompatibility Testing; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Embryonal: Embryonal tumors, including medulloblastoma and ATRT
  Interventions: Diagnostic Test: Tissue, blood, cerebrospinal-spinal fluid
- Glioma, IDH-mutated: IDH-mutated gliomas, including WHO grades 2, 3 and 4
  Interventions: Diagnostic Test: Tissue, blood, cerebrospinal-spinal fluid

INTERVENTIONS:
Diagnostic Test: Tissue, blood, cerebrospinal-spinal fluid — Processing, analysis

SUMMARY:
The treatment of adolescents and young adults (AYA, 15 to 39 years) with malignant intra-axial CNS parenchymal tumors such as IDH-mutated gliomas, medulloblastomas and ependymomas is still not curative in all cases. The tumor biology and clinical needs to diagnose and treat these tumors are comparable across all age groups, so an integrated treatment environment overseen by adult and pediatric neuro-oncology specialists seems promising to leverage synergisms and advance diagnostic and therapeutic development in these tumors. A comprehensive, prospective and integrated biomaterial and imaging-based pipeline for the multi-faceted evaluation of AYAs has not yet been established for AYA patients with brain tumors in Germany. Current diagnostic platforms neglect the integrative processing of data from MRI and FET-PET imaging, radiotherapy plans, tumor tissue, liquid biopsies and clinical data as well as prognostic markers. A prospective AYA pipeline can therefore enable a better understanding of the aforementioned high-risk CNS malignancies and promises clinical advances for AYA patients and the clinical and scientific research landscape.

DETAILED DESCRIPTION:
Objectives: We are conducting a non-interventional study for AYAs with malignant intraaxial CNS parenchymal tumors. All 6 Bavarian BZKF sites are involved in the study. We will collect data on diagnostic and prognostic MRI and FET-PET imaging, quality assurance in radiotherapy and radiotherapy treatment patterns, diagnostic and predictive liquid biopsies from CSF and blood and targeted therapy approaches and integrate them bioinformatically with clinical data.

Work packages: WP01 Prediction of diagnosis by artificial intelligence (AI)-assisted processing of MRI and FET-PET; WP02 Analysis of response and relapse patterns by AI-assisted processing of MRI and FET-PET; WP03 Quality control of radiotherapy planning and patterns-of-care analysis; WP04 Prediction of response, relapse and treatment density using markers identified in liquid biopsies from CSF and blood; WP05 Identification of targets for targeted therapy from paraffin-embedded tissue (FFPE), CSF and blood; WP06 Investigation of clinical patterns and progression (PFS) or WP07 Bioinformatic integration of data to predict PFS, OS and patterns of response, relapse, treatment density and potential molecular targets.

Inclusion criteria: (1) first diagnosis of high-risk CNS tumors including IDHmutated gliomas, medulloblastomas, ependymomas, and other intra-axial primary brain tumors; (2) adolescents and young adults (AYA; 15 to 39 years); (3) Karnofsky status of 60 or higher; (4) multimodality therapy planned at the discretion of the medical professional; (5) expected survival min. 6 months; (6) informed consent by patient and (for patients under 18 years) legal representative; (7) complete material collection expected.

Exclusion criteria: (1) synchronous independent tumor disease, except basal cell carcinoma and carcinoma in situ; (2) participation in interventional clinical trial, except in standard arms of interventional clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. first diagnosis of high-risk CNS tumors including glioma IDHmutated, medulloblastoma, ependymoma and other intra-axial primary brain tumors
2. adolescents and young adults (AYA; 15 to 39 years)
3. Karnofsky status of 60 or higher
4. resection, extended biopsy or stereotactic biopsy with sufficient tissue volume
5. multimodal therapy planned at the discretion of the treating specialist
6. expected survival time of at least 6 months
7. informed consent from the patient or the patient's legal guardian prior to the first study procedure
8. complete material collection expected.

Exclusion Criteria:

1. synchronous independent tumor disease other than basal cell carcinoma and carcinoma in situ
2. participation in interventional clinical trial except in standard arms of interventional clinical trials.

Ages: 15 Years to 39 Years | Sex: All
Age Groups: Child, Adult
Study Population: A total of 72 patients with complete data and biomaterial collection will be recruited into the study, including 36 patients with glioma IDHmutated and 36 patients with pediatric primary intra-axial brain tumors (medulloblastoma, ependymoma, ATRT, others).
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
AI processing of MRI fand PET or diagnosis | March 2026
  Prediction of diagnosis by artificial intelligence (AI)-assisted processing of magnetic resonance imaging (MRI) and Fluorethyltyrosin-Positron Emission Tomography (FET-PET)
AI processing of MRI and PET for evaluation of response and relapse | March 2026
  Analysis of response and relapse patterns by artificial intelligence (AI)-assisted processing of magnetic resonance imaging (MRI) and Fluorethyltyrosin-Positron Emission Tomography (FET-PET)
Quality control analysis in radiotherapy | March 2026
  Quality control of radiotherapy planning and patterns-of-care analysis
Analysis of response in liquid biopsies | March 2026
  Prediction of response using markers detected in liquid biopsies from cerebrospinal fluid and blood
Target molecules in tissue and liquid biopsies | March 2026
  Identification of target molecules for targeted therapy from paraffin-embedded tissue (FFPE), cerebrospinal fluid and blood
Evaluation of progression free survival | March 2026
  Investigation of clinical patterns of response in view of progression free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hau, Prof., Principal Investigator — University Hospital Regensburg

IPD SHARING:
Plan to Share IPD: No
Internal analysis in BZKF network